CLINICAL TRIAL: NCT00881504
Title: A Single-Center, Open-Labeled, Phase II Trial of Modified FOLFOX6 With Bevacizumab in Patients With Advanced Biliary System Carcinoma
Brief Title: A Study of FOLFOX6 With Bevacizumab for Biliary System Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: It was not possible to get insurance companies to cover bevacizumab.
Sponsor: Georgetown University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OX-07-006; 2007-411 (Other: IRB)
Record Dates: First submitted 2009-04-13; First posted 2009-04-15 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-09

CONDITIONS: Biliary Tract Cancer
Keywords: Biliary; Oxaliplatin; Bevacizumab
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Bevacizumab; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- "FOLFOX6" and "Bevacizumab" (Experimental): Intervention = "bevacizumab" in combination with chemotherapy
  Treatment of biliary system carcinoma using "Bevacizumab" in combination with "modified FOLFOX6".
  Interventions: Drug: "Bevacizumab" in combination with "modified FOLFOX6".

INTERVENTIONS:
Drug: "Bevacizumab" in combination with "modified FOLFOX6". — Oxaliplatin 85 mg/m2 IV on Day 1 5-FU: 400 mg/m2 IV bolus on Day 1, followed by 2400 mg/M2 over 46 hours Leucovorin: 400 mg IV Day 1 Bevacizumab: 10 mg/kg IV on Day 1 Repeat cycles every 2 weeks until death, disease progression, unacceptable toxicity, patient refusal, or treatment delay > 4 weeks
  Other Names: Avastin; Eloxatin

SUMMARY:
This study is for patients with biliary tract cancer that has spread and who are not candidates for surgical resection.

The purpose of this research is to determine if bevacizumab can be safely administered with Modified FOLFOX 6 and find out what effects, good and/or bad, this type of treatment has on biliary cancer.

In this study, a combination of chemotherapy, Modified FOLFOX6 and a biologic agent, bevacizumab will be tested.

Subjects on this study will receive chemotherapy and bevacizumab every 2 weeks until their disease gets worse or they are unable to tolerate treatment.

DETAILED DESCRIPTION:
This is a single-center, open labeled, single-arm study in patients with previously untreated unresectable biliary tract cancer. This trial will follow a Simon's two-stage optimal design. For the first stage, 9 patients will be accrued. If none of the 9 patients have controlled disease with mFOLFOX6 in combination with bevacizumab, the combination will be rejected and the trial stopped. However, if at least 1 patient of the 9 (11%) respond to treatment in the first stage, then an additional 15 patients will be entered into the second stage, for a total of 24 patients in the phase II study. If 3 (13%) or more patients respond to therapy, then the combination will be considered for further investigation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of non-resectable adenocarcinoma of the biliary tract, including carcinomas of the gallbladder, the intrahepatic or extrahepatic biliary tract, and ampullary cancer
* Measurable or evaluable disease
* Locally advanced disease that is inoperable ot patients who have had disease recurrence after curative surgical attempt
* Ambulatory with an ECOG performance status of 0-1
* Adequate organ and marrow function
* Must agree to avoid pregnancy prior to study entry and throughout the duration of study participation
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Any prior chemotherapy
* Patients who are receiving other investigational agents
* Patients who have received radiotherapy to more than 25% of their bone marrow for any reason
* Peripheral neuropathy >/= 2
* Known brain metastases, uncontrolled seizure disorder, encephalitis
* Prior history of hypertensive crisis or hypertensive encephalopathy, uncontrolled hypertension,unstable angina, congestive heart failure of New York Heart Association (NYHA) class 2 or greater, left ventricular ejection fraction less than 50%, clinically significant vascular disease, serious cardiac arrhythmia requiring medication, cardiomyopathy
* History of myocardial infarction, unstable angina or stroke/transient ischemic attack (TIA) within 6 months
* History of allergy to oxaliplatin, 5-fluoruracil (5-FU), Leucovorin, or Bevacizumab
* History of intra-abdominal abscess within 4 weeks of study entry, abdominal fistula, gastrointestinal perforation, active peptic ulcer disease, or inflammatory bowel disease
* Evidence of bleeding diathesis or coagulopathy
* Serious non-healing wound, ulcer, or bone fracture
* Major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks of study entry or anticipation of need for major surgery during the course of the study
* Minor surgical procedures such as core biopsies within 7 days before enrollment, chemotherapy port placement within 24 hours
* Patients on full-dose anticoagulants who have out of range international normalized ratio (INR) or active bleeding
* Concurrent malignancy unless the subject has been curatively treated and disease free for >/= 2 years or the cancer was non-melanoma skin cancer or early cervical cancer
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* Known HIV or Hepatitis B or C
* Life expectancy less than 12 weeks
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-06; Primary Completion 2011-02 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John L Marshall, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9 patients were recruited over the course of the study (2009-2011). All were recruited at Georgetown University Medical Center
Groups:
- FOLFOX6 and Bevacizumab: Treatment with modified FOLFOX6 and Bevacizumab
  Modified FOLFOX6 and Bevacizumab: Oxaliplatin 85 mg/m2 IV on Day 1 5-FU: 400 mg/m2 IV bolus on Day 1, followed by 2400 mg/M2 over 46 hours Leucovorin: 400 mg IV Day 1 Bevacizumab: 10 mg/kg IV on Day 1 Repeat cycles every 2 weeks until death, disease progression, unacceptable toxicity, patient refusal, or treatment delay > 4 weeks
Period: Overall Study
Arm/Group | FOLFOX6 and Bevacizumab
Started | 9
Completed | 8
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 3 males; 5 females. Average age, 68.1 years.
Arm/Group | FOLFOX6 and Bevacizumab
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free Survival is defined as the time from randomization (or study initiation) until objective tumor progression or death.
Time Frame: 2 years
Population: Primary outcome of 4 participants out of 8 was undetermined due to several reasons including patient refusal of further follow up.
  Of the 4 patients remaining for analysis, progression free survival of 34, 26.3, 7, and 4.7 weeks was seen.
Measure: Median (Full Range); unit: weeks
Arm/Group | FOLFOX6 and Bevacizumab
Number analyzed (Participants) | 4
weeks | 16.7 [4.7 to 34]

2. Secondary Outcome: Safety and Toxicity
Description: The number of patients who underwent FOLFOX dose reductions as a result of Grade 3 toxicity.
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | FOLFOX6 and Bevacizumab
Number analyzed (Participants) | 8
participants | 3

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | FOLFOX6 and Bevacizumab
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFOX6 and Bevacizumab (N=8)
Perforation of colon (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFOX6 and Bevacizumab (N=8)
anorexia (General disorders) | 4 (4)
hypoalbuminemia (Blood and lymphatic system disorders) | 3 (3)
hypocalcemia (General disorders) | 3 (3)
constipation (Gastrointestinal disorders) | 6 (6)
diarrhea (Gastrointestinal disorders) | 3 (3)
fatigue (General disorders) | 7 (7)
hyperglycemia (Endocrine disorders) | 5 (5)
mucositis/stomitis (General disorders) | 4 (4)
nausea (Gastrointestinal disorders) | 4 (4)
sensory neuropathy (Nervous system disorders) | 6 (6)
low platelet count (Blood and lymphatic system disorders) | 3 (3)
hyponatremia (Gastrointestinal disorders) | 4 (4) — low sodium
vomiting (Gastrointestinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes